CLINICAL TRIAL: NCT07328256
Title: Effects of Post Isometric Relaxation as Compared to Post Isometric Stretching Muscle Energy Technique in the Management of Neck Pain
Brief Title: Effects of Post Isometric Relaxation as Compared to Post Isometric Stretching Muscle Energy Technique in the Management of Neck Pain: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/08
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-10

CONDITIONS: Chronic Neck Pain
Keywords: Subacute neck pain; Neck Muscles; Chronic Neck Pain; Pain Management; Muscle Relaxation; Isometric Contraction
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post Isometric Relaxation (Active Comparator): Post-Isometric Relaxation (PIR) is used for treating muscle tightness or spasms. It involves a sequence of steps that aim to improve flexibility and reduce muscle tension.
  Interventions: Procedure: Post Isometric Relaxation
- Post Isometric Stretching (Experimental): Post-Isometric Stretching (PIS) is a technique used improve flexibility while working on passive tone of the muscle
  Interventions: Procedure: Post Isometric Relaxation; Procedure: Post Isometric Stretching

INTERVENTIONS:
Procedure: Post Isometric Relaxation — All patients were given Trans-Cutaneous Electrical Nerve Stimulation (TENS) in combination with superficial heat for 10 minutes. with a session of 5 days/ week.
  Group A (PIR) : In this group, participants performed 3-5 rounds of post-isometric relaxation (PIR). Each round involved contracting the target muscle at 30-50% strength for 7-10 seconds, resting for 5 seconds .
Procedure: Post Isometric Stretching — All patients were given Trans-Cutaneous Electrical Nerve Stimulation (TENS) in combination with superficial heat for 10 minutes. with a session of 5 days/ week.Group B (PIS) : In this group participants performed 3-5 rounds of post-isometric relaxation (PIR), which is then followed by a stretch of the same muscle to its new range of motion. Followed by rest of 5 seconds, and then stretching the muscle and holding the stretch for 10-60 seconds
  Arms: Post Isometric Stretching

SUMMARY:
This study aims to compare the effects of post-isometric relaxation (PIR) and post isometric stretching (PIS) techniques on reducing neck pain, improving range of motion, and decreasing neck disability in individuals with neck pain. A randomized controlled trial will be conducted with 50 participants, who will be randomly assigned to one of two groups: one receiving PIR and the other receiving PIS. A single-blind method will be used, meaning the participants will not know which group they belong to. Participants will be selected based on specific criteria related to neck pain and will then be randomly allocated to the PIR or PIS group. Initially, all participants will receive two standard treatments: Transcutaneous Electrical Nerve Stimulation (TENS) and hot pack application. After these treatments, one group will undergo post-isometric relaxation (PIR), which involves 3-5 repetitions of muscle contraction and relaxation, conducted over five consecutive sessions. The other group will receive post-isometric stretching (PIS), which involves stretching after muscle contraction and relaxation, also administered over five consecutive sessions. At the end of the intervention, pain, range of motion, and neck disability will be measured. Pain will be assessed using a standardised pain scale, range of motion will be measured with a goniometer or other appropriate tools, and neck disability will be evaluated using the Neck Disability Index (NDI). Statistical analysis will be performed to compare the effectiveness of PIR and PIS in terms of pain reduction, range of motion improvement, and decreased neck disability.

DETAILED DESCRIPTION:
Neck pain is one of the most prevalent musculoskeletal complaints among young adults, with studies reporting a prevalence of up to 75.7%, making it the fourth leading cause of disability worldwide. Research suggests that weak cervical musculature, reduced muscle-to-bodyweight ratios, and imbalances in muscle strength are key contributors to neck pain and associated disability. Muscle Energy Techniques (METs), particularly Post-Isometric Relaxation (PIR) and Post-Isometric Stretching (PIS), have been widely used to address these issues. PIR involves gentle isometric contractions followed by muscle relaxation and is effective for managing active muscle tone, making it suitable for acute conditions. However, it lacks a stretching component to target passive tone. PIS adds a post-contraction stretch, potentially addressing both active and passive tone, but may cause discomfort in sensitive individuals. While both techniques have shown positive outcomes in reducing pain and improving function, limited research directly compares their effectiveness. Therefore, this study aims to compare PIR and PIS in terms of pain relief, cervical range of motion, and functional improvement in individuals with mechanical neck pain.

According to M.Osama et al in 2020 a study was conducted to compared autogenic inhibition (AI) and reciprocal inhibition (RI) muscle energy techniques (MET) to static stretching (SS) for managing mechanical neck pain. Both AI-MET and RI-MET outperformed SS in enhancing isometric strength, with no adverse effects observed. The findings highlight AI-MET's superiority and support its use in neck pain rehabilitation.

Another study was conducted by Osama M 2024, 78 participants a randomized trial concluded that Muscle and Movement specific PIR is effective in improving neck pain, disability and ROM. Dudonienė V et al preformed a study in 2024 that aimed to investigate the 3 effectiveness of post-isometric relaxation (PIR) compared to self-stretching (SS) in working-age individuals with chronic non-specific neck pain. Result showed PIR group achieved lower pain intensity, greater neck extension ROM and lower neck disability index compared to the SS group.

A study conducted in 2022 investigates the effects of post-isometric relaxation (PIR) versus myofascial release therapy on non-specific neck pain management. Results showed that the PIR group had significant improvements in pain (measured by VAS), disability (NDI), cervical extension, and social QoL compared to the MFR group.

Another study investigated the effectiveness of post isometric relaxation (PIR) combined with traditional physical therapy for treating chronic mechanical neck pain compared to traditional therapy alone. Results showed significant reductions in pain and increases in cervical range of motion (ROM) for group adding PIR to conventional therapy.

The study compares the effectiveness of post-isometric relaxation (PIR) and passive neck retraction mobilization (PNRM) in treating nonspecific neck pain. This study suggests that PIR to be a more effective treatment option for nonspecific neck discomfort.

ELIGIBILITY:
Inclusion Criteria: • Age ranging from 19-44 years old

* Both gender
* With sub-acute or chronic neck pain for at least 4 to 12 weeks
* Pain intensity on NPRS ranging 4-8
* Limitation on neck movement

Exclusion Criteria:

* • Positive history of fracture

  * Surgery in the cervical region
  * Any sort of physical trauma in the cervical region in the last 12 months
  * Thoracic Outlet syndrome
  * Cervical radiculopathy
  * Cervical myelopathy
  * Cervical spondylosis
  * Cervical syringomyelia
  * Any systemic disorder including malignancy or inflammatory and rheumatic disorders
  * Infection
  * Vascular syndromes such as vertebrobasilar insufficiency (VBI).

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 1 week
  The Visual Analog Scale (VAS) will be used to measure the intensity of neck pain before and after the intervention. Participants will mark their level of pain on a 100 mm horizontal line, where:
  0 mm indicates "no pain", and 100 mm indicates "the worst imaginable pain".
Cervical range of motion | 1 week
  A universal goniometer will be used to assess cervical spine mobility in the following directions:
  Flexion Extension Lateral Flexion (Right and Left) Rotation (Right and Left) ROM will be recorded in degrees.
Functional Disability | 1 week
  The Neck Disability Index (NDI) will be used to assess functional impairment related to neck pain. It is a self-administered questionnaire consisting of 10 sections, including pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation.
  Each section is scored from 0 to 5, with higher total scores indicating greater disability. The NDI is a validated, open-access tool commonly used in research to measure changes in disability levels pre- and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: FUI, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Punjab Province, Pakistan